CLINICAL TRIAL: NCT07228923
Title: Evaluation of a Theory Informed Intervention to Reduce Hazardous Alcohol Consumption Among Treatment Seeking Smokers
Brief Title: Development and Evaluation of a Theory and Evidence-based Intervention to Reduce Hazardous Alcohol Consumption Among Treatment Seeking Smokers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCP-196026
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Alcohol Misuse
Keywords: Smoking Cessation; Alcohol; Brief Intervention; SBIRT
MeSH Terms: conditions — Smoking Cessation | interventions — Ethanol; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient Portal Prompt (Experimental): Brief Alcohol Intervention
  Interventions: Behavioral: Brief alcohol intervention

INTERVENTIONS:
Behavioral: Brief alcohol intervention — The intervention is a prompt that that appears as an alert message in the patient portal, recommending the alcohol intervention.

SUMMARY:
This study will evaluate the implementation of a fully automated, direct-to-patient digital alcohol intervention embedded within the STOP Program's patient portal. The STOP Program is a large-scale, population-based smoking cessation initiative operating in over 300 primary care settings across Ontario. It provides free nicotine replacement therapy and behavioural support through a digital portal that facilitates patient self-enrollment and systematic data collection. As part of this study, patients who score ≥8 on the AUDIT-C will be offered the opportunity to view a brief intervention (BI). Those with an AUDIT-C score ≥10 will receive a cautionary message along with tailored content designed to help reduce hazardous drinking.

The intervention was developed based on a rapid review (PROSPERO: CRD42023445492) and a Delphi consensus process using the Behaviour Change Techniques Taxonomy V1. Key components include personalized feedback, normative comparisons, reflective prompts, and actionable behaviour change strategies. For patients scoring above a clinical threshold, additional messaging encourages caution regarding abrupt cessation and suggests consulting a healthcare provider.

Our primary outcome is acceptance of the new online resource.

ELIGIBILITY:
Inclusion Criteria:

* seeking treatment for smoking cessation
* enrolling via the patient self-serve portal
* AUDIT-10 score of 8 or higher

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
overall acceptance rate | Data will be collected at baseline

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-10-20): https://cdn.clinicaltrials.gov/large-docs/23/NCT07228923/SAP_000.pdf